CLINICAL TRIAL: NCT04954313
Title: Baseline Oral Health Study: UnCoVer the Connections to General Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-1453; CRO-2020-03-VERILY-LK (Other: Verily)
Record Dates: First submitted 2021-06-22; First posted 2021-07-08 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Diabetes Type 2
Keywords: Oral health
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and all sub-investigators will make every effort to remain blinded as to the subject regimen. Periodontal treatment throughout the Study will be provided only by experienced general dentists, periodontists or dental hygienists who are licensed, trained and calibrated prior to the start of the study. In order to maintain examiner blinding throughout the study, the treatment provider will be a person other than the dental examiner and will exclusively provide treatment and not participate in patient assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): The Treatment Group will receive the same periodontal treatment in addition to having subgingival chlorhexidine irrigation. All subjects will also complete a set of questionnaires (PANAS & PMT) using an online form. A subset of 50 subjects from each group will be randomly selected to have oral images captured using an intra-oral scanner at Baseline and a subset of follow-up visits. Additionally, subjects in the Treatment Group will also receive brief behavioral advice from dental professionals focusing mainly on motivation and acknowledgement.
  Interventions: Drug: Subgingival chlorhexidine irrigation; Other: Dental Supplies; Other: Periodonal Treatment
- Control Group (Active Comparator): The Control Group will receive an initial periodontal treatment consisting of a pre-procedural rinse and scaling & root planning (SRP).
  Subjects in the Control Group will receive no products during the course of the study. They will receive a commercial connected toothbrush, toothpaste, mouthwash, proxabrush, and floss at the end of the study. Subjects will be scheduled to receive flow mediated dilation (FMD) and carotid intima media thickness (IMT) measurements prior to Baseline and approximately 4 weeks after their Baseline visit.
  Interventions: Other: Periodonal Treatment

INTERVENTIONS:
Drug: Subgingival chlorhexidine irrigation — The dose information for the Chlorhexidine gluconate will be 0.12% with 1 mL in each dental pocket at a frequency of every 3 months for the duration of the study (18 months).
  Arms: Treatment Group
Other: Dental Supplies — Subjects in the Treatment Group will receive a commercial electric toothbrush (Colgate hum), toothpaste (Colgate Renewal), mouthwash (Colgate Zero), proxabrush (Colgate), and floss (Colgate Palmolive brand) to be used at home along with instructions on their use. Brush heads for the electric toothbrush will be replaced every 3 months and products (toothpaste, mouthwash, proxabrush, and floss) will be replenished at every site visit.
  Arms: Treatment Group
Other: Periodonal Treatment — Initial periodontal treatment consisting of a pre-procedural rinse and scaling & root planing (SRP).

SUMMARY:
Purpose: The Baseline Oral Health Health Study is a randomized controlled trial to evaluate the impact of regular, professional non-surgical Intensive Periodontal Therapy (scaling and root planing and optimal oral hygiene with associated professional oral health behavior advice ), on oral health as well as whether such effects are associated with corresponding changes to biomarkers characterizing systemic health.

Participants: The Baseline Oral Health Study will enroll approximately 200 participants in the study with approximately 100 participants each within the Control Group and the Treatment Group. The study population will be recruited from the Project Baseline Health Study participants in the North Carolina region and may be expanded to include subjects recruited from University of North Carolina (UNC) if the initial screening from Project Baseline Health Study pool of participants in the North Carolina region does not fulfill study enrollment powering.

Procedures (methods): The study population will be recruited from Project Baseline Health Study participants. The Project Baseline Health Study is a longitudinal cohort study which characterizes participants across clinical, molecular, imaging, sensor, self-reported, behavioral, psychological, environmental, or other health-related measurements from onsite and/or remote visits, continuous monitoring through sensor technology, and regular engagement via an online portal, and mobile app. The study population will be recruited from Project Baseline Health Study participants diagnosed with cardiovascular disease and/or type 2 diabetes mellitus (including prediabetes) and eligible for periodontal intervention. The study will use dental centers and an experienced dental team to manage the oral care provided in this study.

DETAILED DESCRIPTION:
The Baseline Oral Health Health Study is a randomized controlled trial to evaluate the impact of regular, professional non-surgical Intensive Periodontal Therapy (scaling and root planing and optimal oral hygiene with associated professional oral health behavior advice ), on oral health as well as whether such effects are associated with corresponding changes to biomarkers characterizing systemic health. The study will be conducted in partnership with Verily and the Project Baseline Team, Colgate, and the University of North Carolina. The study population will be recruited from Project Baseline Health Study participants. The Project Baseline Health Study is a longitudinal cohort study which characterizes participants across clinical, molecular, imaging, sensor, self-reported, behavioral, psychological, environmental, or other health-related measurements from onsite and/or remote visits, continuous monitoring through sensor technology, and regular engagement via an online portal, and mobile app.

The study population will be recruited from Project Baseline Health Study participants diagnosed with cardiovascular disease and/or type 2 diabetes mellitus (including prediabetes) and eligible for periodontal intervention. The study will use dental centers and an experienced dental team to manage the oral care provided in this study.

ELIGIBILITY:
Inclusion Criteria:

* At least eighteen (18) years of age but not older than seventy (70) years of age at the time of screening
* Able to speak and read English
* Has at least 16 teeth present.
* Able to consent, follow an outpatient protocol, and is available by telephone
* Has either moderate (stage II) or severe (stage III) periodontitis:

  * Stage II - Interdental clinical attachment level (CAL) at the site of greatest loss = 3 to 4mm with maximum probing depth ≤ 5mm
  * Stage III - Interdental CAL at the site of greatest loss ≥ 5mm, probing depth (PD)≥ 6mm, and radiographic bone loss (vertical bone loss ≥ 3mm)
* Has at least one of the following indicators of cardiometabolic disease in the following range:

  * Type 2 diabetes: 9% ≥ HbA1c ≥ 6.5% OR Prediabetes: 6.4%≥ HbA1c ≥ 5.7% OR
  * Cardiovascular Disease (CVD):

    * Medical history of Myocardial Infarction, Coronary Artery Disease or stroke
* Access to Apple (iOS) devices or Android devices with appropriate versions to be compatible with the applications to complete study procedures.
* Females of childbearing capacity must be willing to have pregnancy test

Exclusion Criteria:

* Individuals who exhibit gross oral pathology
* Presenting oral manifestations of systemic diseases (e.g. pemphigus, pemphigoid, lupus)
* Presence of any acute or chronic systemic infection as determined by the clinician
* Periodontal treatment performed within 6 months prior to study start
* Refusal to extract hopeless teeth identified as determined by the clinician at the screening visit.
* Participating in any other interventional cardiometabolic or Oral Health study
* Individuals currently undergoing any type of orthodontic treatment (e.g. aligners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroja Voruganti, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - UNC Nutrition Research Institute, Kannapolis, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 786 participants who signed informed consent, 194 completed the required assessments, and remained eligible. Of the 194 eligible participants, 39 declined to be randomized. Of the 155 randomized participants, two did not continue following randomization and did not receive any exposure to a study intervention.
Groups:
- Control Group: The Control Group will receive an initial periodontal treatment consisting of a pre-procedural rinse and scaling & root planning (SRP).
  Subjects in the Control Group will receive no products during the course of the study. They will receive a commercial connected toothbrush, toothpaste, mouthwash, proxabrush, and floss at the end of the study. Subjects will be scheduled to receive flow mediated dilation (FMD) and carotid intima media thickness (IMT) measurements prior to Baseline and approximately 4 weeks after their Baseline visit.
  Periodontal Treatment: Initial periodontal treatment consisting of a pre-procedural rinse and scaling & root planing (SRP).
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 73 | 82
Completed T0 (Day 0) | 73 | 80
Completed T1 (Day 90) | 65 | 70
Completed T2 (Day 180) | 61 | 65
Completed T3 (Day 270) | 56 | 57
Completed T4 (Day 360) | 54 | 56
Completed | 53 | 54
Not Completed | 20 | 28
Not completed — Lost to Follow-up | 6 | 12
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 11 | 13
Not completed — Physician Decision | 0 | 1
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: two participants withdrew between randomization and first intervention
Groups:
- Control Group: The Control Group will receive an initial periodontal treatment consisting of a pre-procedural rinse and scaling & root planning (SRP).
  Subjects in the Control Group will receive no products during the course of the study. They will receive a commercial connected toothbrush, toothpaste, mouthwash, proxabrush, and floss at the end of the study. Subjects will be scheduled to receive flow mediated dilation (FMD) and carotid intima media thickness (IMT) measurements prior to Baseline and approximately 4 weeks after their Baseline visit.
  Periodonal Treatment: Initial periodontal treatment consisting of a pre-procedural rinse and scaling & root planing (SRP).
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 73 | 80 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 72 | 138
  >=65 years | 7 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 89
  Male | 31 | 33 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 41 | 77
  White | 30 | 33 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Diabetes/pre-diabetes [Count of Participants; unit: Participants] — Prediabetes/diabetes defined as HbA1c at screening >=5.7 Population: HbA1c was measured at screening for classification. For one participant, HbA1c at screening was not recorded and classification was based on HbA1c measured at T0 (day 0). For two participants, HbA1c was not recorded at screening not recorded at T0, and no prediabetes/diabetes classification was made.
  Participants
    Prediabetes/diabetes ( HbA1c >=5.7 at screening) | 57 | 64 | 121
    Non-prediabetes/non-diabetes ( HbA1c < 5.7 at screening) | 16 | 14 | 30
    Uncategorized (HbA1c not recorded at screening or T0) | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Impact of Treatment on Change in Oral Health Measures
Description: The impact of treatment on oral health measures, will be performed using generalized estimating equations (GEE) methods. Longitudinal outcomes in the Treated vs. Control groups will be compared and will include all subjects who were randomized and their data from visits T1 - T4 based on intent-to-treat (ITT) group assignment. Periodontal probing depths (mm) will be measured per sextant. Whole-mouth mean probing depths will be used as a measure of oral health.
Time Frame: Comparing T1 (day 90) and T4 (day 360)
Population: Data include imputation. Predictions based on linear mixed models were used for imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters (probing depth difference)
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 73 | 80
millimeters (probing depth difference) | 0.186 [0.0863 to 0.285] | 0.190 [0.0737 to 0.306]
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; Difference in change from T1 to T4 between the control and treatment groups was quantified using a difference-in-difference estimate; Test type: Superiority; p = 0.957, Generalized Estimating Equations — p values are presented without adjustment for multiple hypotheses; difference in difference of LSM = -0.00419, 95% CI 2-sided [-0.157 to 0.149] — Change from T1 to T4 in the control group compared to the treatment group

2. Primary Outcome: Association Between Changes in Oral Health (Probing Depth) and Changes in Systemic Health (HbA1c)
Description: The association between changes in oral health and changes in systemic health, will be evaluated using correlation analysis. Periodontal probing depths (mm) will be measured per sextant. Whole-mouth mean probing depths will be used as a measure of oral health. The correlation between % change in whole-mouth mean probing depth and % change in HbA1c will be determined in subjects with prediabetes or type 2 diabetes at screening.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants meeting the following criteria: (1) HbA1c data was available at T0 and T4 time points, (2) probing depth data was available at T0 and T4 time points, and (3) screening HbA1c >= 5.7 (if screening value was not available, T0 value of HbA1c >= 5.7 was used as proxy).
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 38 | 46
Pearson correlation coefficient | -0.093 (0.379) | -0.282 (0.5123)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; This outcome used linear regression to test the hypothesis of a correlation between change in probing depth and change in HbA1c in diabetic/prediabetic participants between timepoints T4 and T0; Test type: Superiority; p = 0.0378, Regression, Linear

3. Primary Outcome: Association Between Changes in Oral Health and Changes in Systemic Health (Flow-mediated Dilation)
Description: The association between changes in oral health and changes in systemic health, will be evaluated using correlation analysis. Periodontal probing depths (mm) will be measured per sextant. Whole-mouth mean probing depths will be used as a measure of oral health. The correlation between % change in whole-mouth mean probing depth and change in flow-mediated dilation will be calculated.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants meeting the following criteria: (1) flow mediated dilation data was available at T0 and T4 time points, (2) probing depth data was available at T0 and T4 time points.
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 46 | 49
Pearson correlation coefficient | -0.0528 (0.3635) | 0.006 (0.5227)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; This outcome used linear regression to test the hypothesis of a correlation between change in probing depth and change in flow mediated dilation between timepoints T4 and T0; Test type: Superiority; p = 0.4735, Regression, Linear

4. Secondary Outcome: Change in Emotional Wellbeing
Description: Emotional wellbeing will be evaluated through the use of PANAS (Positive Affect and Negative Affect Scales). PANAS consists of 10 positive and 10 negative valence word items. Items are rated by the participant to indicate their assessment of how they are feeling about this item "right now" on a scale of 1(slightly) or not at all through 5 (extremely). 10 of of the items form a positive affect subscale, in which a higher score indicates increased positive affect, with a subscale range of 10 to 50. 10 of the items form a negative affect subscale, in which a higher score indicates more negative affect, with a subscale range of 10 to 50. This outcome measure is change in the 10 item positive affect subscale.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants who completed the survey at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 16 | 15
scores on a scale | 1.25 (6.93) | -0.6 (7.09)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for change of emotional wellbeing as measured by positive affect subscore from PANAS survey, from baseline (T0) to day 360 (T4) and is calculated as (PANAS@T4 - PANAS@T0) for each participant who completed the survey at T0 and T4; Test type: Superiority; p = 0.469, t-test, 2 sided

5. Secondary Outcome: Change in Beliefs About Periodontal Disease
Description: Beliefs about periodontal disease will be evaluated through the use of a Protective Motivation Theory (PMT) survey. PMT surveys assess an individual's motivation to adopt protective health behaviors by focusing on specific cognitive processes. This survey includes 7 statements related to opinions on periodontal disease and treatment (e.g., "Periodontal disease worries me," "Adhering to my periodontal treatment instructions over the next weeks will improve my oral health"). Each survey item is scored from 1 to 10 with 1 being "not at all" to 10 being "extremely so." Higher values indicate stronger agreement with the survey statements. Reported outcome measures represent total survey scores (range from 7 to 70).
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants who completed the survey at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 16 | 15
scores on a scale | 2.56 (8.75) | -0.60 (4.47)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for beliefs about periodontal care as measured by PMT survey from baseline (T0) to day 360 (T4) and is calculated as (PMT_sum@T4 - PMT_sum@T0) for each participant with measurement data in each group; Test type: Superiority; p = 0.220, t-test, 2 sided

6. Secondary Outcome: Change in Bleeding on Probing
Description: Whole-mouth mean of tooth-specific dichotomic response (bleeding = 1, no bleeding = 0) after probing the gingival sulcus.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants who received dental assessment at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 54 | 56
scores on a scale | -0.109 (0.188) | -0.212 (0.236)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for bleeding on dental probing of the gingival sulcus from baseline (T0) to day 360 (T4) and is calculated as (BOP@T4 - BOP@T0) as scored by index (bleeding = 1 and no bleeding = 0), and averaged across the mouth for each participant with measurement data in each group; Test type: Superiority; p = 0.014, t-test, 2 sided

7. Secondary Outcome: Change in Gingival Index
Description: The gingival index will be scored on three facial surfaces (distofacial, facial, mesiofacial) and three lingual surfaces (distolingual, lingual, mesiolingual). Areas are examined by placing the periodontal probe under the gingival margin at approximately 1mm deep and sweeping the probe from the distal surface to the mesial surface in quadrants I and IV and mesial to the distal surface in quadrants II and III. After each quadrant is swept, calls are made based on gingival inflammation and the presence or absence of bleeding according to criteria which range from 0 to 3. Loe and Silness Gingival Index (GI); scale: 0 = normal gingiva, 1 = mild inflammation, 2 = moderate inflammation, 3 = severe inflammation. For this Outcome Measure, less inflammation (lower number) correlates with better outcome. Reported outcome measure is whole-mouth mean value (six surfaces of each tooth), with a range of 0 to 3.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants who received dental assessment at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 54 | 56
scores on a scale | -0.154 (0.47) | -0.379 (0.559)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for change of gingival index from baseline (T0) to day 360 (T4) and is calculated as (GI@T4 - GI@T0) mean across all teeth for each participant with measurement data in each group; Test type: Superiority; p = 0.025, t-test, 2 sided

8. Secondary Outcome: Percent Change in Clinical Attachment Level (CAL)
Description: Percent change of whole-mouth mean clinical attachment level (CAL, defined as measured pocket depth - gingival margin, for each site). Percent change calculated as (CAL@T4 - CAL@T0)/CAL@T0.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants who received dental assessment at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 54 | 56
% change | -0.31 (22.2) | 0.90 (25.2)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for percent change of clinical attachment level (gingival margin relative to crown margin) from baseline (T0) to day 360 (T4) and is calculated as (CAL@T4 - CAL@T0)/CAL@T0 (mean across teeth) for each participant with measurement data in each group; Test type: Superiority; p = 0.79, t-test, 2 sided

9. Secondary Outcome: Change in Dental Plaque Index
Description: Change of digitally measured interdental plaque area. Full mouth plaque assessment shall be assessed using the UNC Modified Plaque Index (Greene and Vermillion). Plaque scores shall be visually assessed at 6 sites per tooth (distobuccal, buccal, mesiobuccal and distolingual, lingual, mesiolingual surfaces) on a scale of 0-3. Scores are the following: 0 =No debris or stain present on the clinical crown; 1 =Soft debris covering not more than 1/3 of the clinical crown (cervical 3rd), or presence of extrinsic stains without other debris regardless of surface area covered; 2 =Soft debris covering more than 1/3, but not more than 2/3 (middle 3rd) of the clinical crown; 3 =Soft debris covering more than 2/3 of the clinical crown. Reported outcome measure is calculated as whole-mouth mean (mean of each site at each tooth) with a range of 0 to 3.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants who received dental assessment at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 54 | 55
scores on a scale | -0.090 (0.579) | -0.181 (0.537)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for dental plaque as assessed by plaque index (scored from 0 to 3) from baseline (T0) to day 360 (T4) and is calculated as (PI@T4 - PI@T0) for each participant with measurement data in each group; Test type: Superiority; p = 0.394, t-test, 2 sided

10. Secondary Outcome: Change in Flow-mediated Dilation
Description: Change of flow mediated dilation. Ultrasound images of the right brachial artery and Doppler measures of arterial flow will be acquired before and after reactive hyperemia is induced by inflating a pneumatic occlusion cuff placed around the lower arm. FMD will be calculated as the percent change in arterial diameter from baseline.
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Some participants did not have FMD measured at T0 and/or T4 and are not included in the T4-T0 comparison. Missing data arises from a combination of participant withdrawal/loss to followup and poor ultrasound data quality.
Measure: Mean (Standard Deviation); unit: % change
Groups:
- Control Group: The Control Group will receive an initial periodontal treatment consisting of a pre-procedural rinse and scaling & root planning (SRP).
  Subjects in the Control Group will receive no products during the course of the study. They will receive a commercial connected toothbrush, toothpaste, mouthwash, proxabrush, and floss at the end of the study.
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 46 | 49
% change | -0.488 (4.97) | 0.45 (4.23)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for difference in flow-mediated dilation (FMD) from baseline (T0) to day 360 (T4) and is calculated as (FMD@T4 - FMD@T0) for each participant with measurement data in each group. FMD is percent change and the comparison of FMD at two timepoints is accomplished by subtraction; Test type: Superiority; p = 0.323, t-test, 2 sided

11. Secondary Outcome: Percent Change in Glycated Hemoglobin (HbA1c) (Prediabetic and Type 2 Diabetic Cohorts)
Description: Percent change of HbA1c (% glycated) from day 0 to day 360 [(HbA1c@T4 - HbA1c@T0) / HbA1c@T0] in the prediabetic and diabetic cohorts (HbA1c >= 5.7 at screening)
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants meeting the following criteria: (1) biomarker data was available at T0 and T4 time points and (2) screening HbA1c >= 5.7 (if screening value was not available, T0 value of HbA1c >= 5.7 was used as proxy).
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 38 | 46
% change | -0.99 (2.21) | -0.65 (1.92)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for percent change of HbA1c from baseline (T0) to day 360 (T4) and is calculated as (HbA1c@T4 - HbA1c@T0) / HbA1c@T0 for each participant with measurement data in each group; Test type: Superiority; p = 0.464, t-test, 2 sided

12. Secondary Outcome: Percent Change in Carotid Intima Media Thickness (IMT)
Description: Percent change of IMT. Longitudinal ultrasound images of the distal 1 cm segments of the right and left common carotid arteries, carotid bulbs, and internal carotid arteries will be acquired. IMT will be measured as the distance between luminal-intimal interface and medial-adventitial interface. Mean IMT will be calculated as the average of all measurements; mean maximum IMT will be calculated as the average of maximum wall thicknesses for each of the regions.
  Percent change of IMT (mm) from day 0 to day 360 is calculated as (IMT@T4 - IMT@T0) / IMT@T0]
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Some participants are missing measurement data at either T0 or T4 timepoints, precluding calculation of T0 to T4 percent change. Missing data arises from a combination of participant withdrawal/loss to followup and poor ultrasound data quality.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 46 | 44
% change | 2.76 (14.9) | 3.48 (18.1)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for percent change of IMT thickness from baseline (T0) to day 360 (T4) and is calculated as (IMT@T4 - IMT@T0) / IMT@T0 for each participant with measurement data in each group; Test type: Superiority; p = 0.838, t-test, 2 sided

13. Secondary Outcome: Percent Change of High Sensitivity C-reactive Protein (Hs-CRP)
Description: Percent change of hs-CRP (mg/dL) from day 0 to day 360 [(CRP@T4 - CRP@T0) / CRP@T0]
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants for whom biomarker data was available at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 51 | 52
% change | -8.56 (70.4) | 21.8 (171)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for percent change of C-reactive protein from baseline (T0) to day 360 (T4) and is calculated as (CRP@T4 - CRP@T0) / CRP@T0 for each participant with measurement data in each group; Test type: Superiority; p = 0.242, t-test, 2 sided

14. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change of total cholesterol (mg/dL) from day 0 to day 360 [(tchol@T4 - tchol@T0) / tchol@T0]
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants for whom biomarker data was available at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 50 | 52
% change | -0.0554 (18.0) | -0.710 (16.2)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for percent change of total cholesterol from baseline (T0) to day 360 (T4) and is calculated as (tchol@T4 - tchol@T0) / tchol@T0 for each participant with measurement data in each group; Test type: Superiority; p = 0.847, t-test, 2 sided

15. Secondary Outcome: Percent Change in Low Density Lipoprotein (LDL) Cholesterol
Description: Percent change of low density lipoproteins (LDL) cholesterol (mg/dL) from day 0 to day 360 [(LDL@T4 - LDL@T0) / LDL@T0]
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants for whom biomarker data was available at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 50 | 51
% change | 2.63 (35.1) | -0.033 (26.0)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for percent change of LDL from baseline (T0) to day 360 (T4) and is calculated as (LDL@T4 - LDL@T0) / LDL@T0 for each participant with measurement data in each group; Test type: Superiority; p = 0.666, t-test, 2 sided

16. Secondary Outcome: Percent Change in Triglycerides
Description: Percent change of triglycerides (mg/dL) from day 0 to day 360 [(trig@T4 - trig@T0) / trig@T0]
Time Frame: Comparing T0 (day 0) and T4 (day 360)
Population: Analysis population includes only participants for whom biomarker data was available at T0 and T4 time points.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 44 | 48
% change | -2.86 (19.3) | -1.52 (21.9)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; The analysis tests the hypothesis that there will be a difference between control and treatment groups for percent change of triglycerides from baseline (T0) to day 360 (T4) and is calculated as (trig@T4 - trig@T0) / trig@T0 for each participant with measurement data in each group; Test type: Superiority; p = 0.758, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From T0 (day 0) through the end of study, up to 15 months
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 1/73 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/73 | 0/80
Other Adverse Events (participants affected / at risk) | 0/73 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=73) | Treatment Group (N=80)
Pancreatitis (Gastrointestinal disorders) | 1 | 0 — participant was a no-show for several scheduled visits and later reported hospitalization for pancreatitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT04954313/Prot_SAP_000.pdf